CLINICAL TRIAL: NCT01643460
Title: Endoscopic Ultrasound (EUS)-Guided Ablation of Pancreatic Cysts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John DeWitt, Director Endoscopic Ultrasound, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0812-57
Record Dates: First submitted 2012-06-28; First posted 2012-07-18 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Pancreatic Cyst; Pancreatic Intraductal Papillary-Mucinous Neoplasm; Cystadenoma, Mucinous; Papillary Mucinous Cystadenoma, Borderline Malignancy
Keywords: Intraductal papillary mucinous neoplasms (IPMNs); Mucinous cystadenomas [MCN]); Invasive IPMNs or mucinous cystadenocarcinomas) tumors
MeSH Terms: conditions — Pancreatic Cyst; Pancreatic Intraductal Neoplasms; Cystadenoma, Mucinous; Cystadenocarcinoma, Mucinous; Neoplasms | interventions — Ethanol; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 98% Ethanol with Paclitaxel injection (Experimental)
  Interventions: Procedure: 98% Ethanol & Paclitaxel injection

INTERVENTIONS:
Procedure: 98% Ethanol & Paclitaxel injection — Pancreatic cyst injection via Endoscopic Ultrasound (EUS)of 98% Ethanol with Paclitaxel (dose determined in relation to cyst size & amount of fluid aspirated from the cyst.
  Other Names: Pancreatic cyst injection of Paclitaxel.

SUMMARY:
The purpose of this study is to track outcomes and complications of patients at IUMC referred by physicians for EUS-guided pancreatic cyst ablation. This information is essential in order to disseminate future published information to physicians about this technique. A database will be created to track these patients undergoing an already scheduled/planned procedure. Phone calls at selected intervals will be made following the procedure to track any complications that occur

DETAILED DESCRIPTION:
Pancreatic cysts represent a wide spectrum of lesions. Many cysts are uniformly benign (pseudocysts) or have negligible malignant potential (serous cystadenomas). However, others represent premalignant (i.e. intraductal papillary mucinous neoplasms (IPMNs) or mucinous cystadenomas [MCN]), or malignant (i.e. invasive IPMNs or mucinous cystadenocarcinomas) tumors. Management of pancreatic cysts is challenging but surgery is generally recommended for cysts that are symptomatic, premalignant (except possibly branch duct IPMNs) or demonstrate malignancy by imaging features and/or biopsy. However, even in experienced hospitals, surgical resection or enucleation of pancreatic cystic tumors is associated with significant perioperative morbidity and mortality rates of 20-40% and up to 2%, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred between January 2009 and February 2016 to EUS at IUMC for pancreatic cyst ablation and with no contraindications for anticipated safe and successful performance of the procedure.
2. Patient at least 18 years of age.

Exclusion Criteria:

1. Investigator deems cyst does not meet safety or need for cyst ablation.
2. Subject not competent to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-09; Primary Completion 2020-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Cyst resolution | 6 months
  1. Patients will undergo EUS-guided cyst ablation with ethanol +/- paclitaxel as indicated for their scheduled procedure. 2. Patients will return 3 months after initial ablation for a repeat EUS, and ablation will be repeated if cyst size is >10mm in diameter. 3. CT or MRI imaging will be performed 3 months after the second procedure to assess for cyst resolution.

CONTACTS AND LOCATIONS:
Overall Officials: John M. DeWitt, MD, Principal Investigator — Indiana University Hospital, Indianapolis, IN 46202
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Kim KH, McGreevy K, La Fortune K, Cramer H, DeWitt J. Sonographic and cyst fluid cytologic changes after EUS-guided pancreatic cyst ablation. Gastrointest Endosc. 2017 Jun;85(6):1233-1242. doi: 10.1016/j.gie.2016.09.011. Epub 2016 Sep 17. PMID 27650271
- [Derived] DeWitt JM, Al-Haddad M, Sherman S, LeBlanc J, Schmidt CM, Sandrasegaran K, Finkelstein SD. Alterations in cyst fluid genetics following endoscopic ultrasound-guided pancreatic cyst ablation with ethanol and paclitaxel. Endoscopy. 2014 Jun;46(6):457-64. doi: 10.1055/s-0034-1365496. Epub 2014 Apr 25. PMID 24770971